CLINICAL TRIAL: NCT07111533
Title: Autogenous Periosteal Pedicle Graft Versus Pericardium Membrane in Management of Periodontal Intrabony Defects in Stage III Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Walaa Ahmed Abd Elaziz Hassanien, Demonstrator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPG vs CM in periodontitis ttt
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis (Stage 3)
MeSH Terms: conditions — Periodontitis | interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Open Flap Debridement (OFD) with autogenous Periosteal Pedicle Graft (PPG) and Bone graft). (Active Comparator): ● In Group I , OFD will be performed, then a bone graft will be packed into the defect and autogenous PPG will be adapted for defect coverage as an autogenous membrane for GTR.
  Interventions: Procedure: Open Flap Debridement (OFD); Procedure: Bone Graft; Procedure: Autogenous Periosteal Pedicle Graft (PPG)
- Group II (Open Flap Debridement (OFD) with Pericardium membrane and Bone graft). (Active Comparator): ● In Group II , OFD will be performed, then a bone graft will be packed into the defect and a pericardium membrane was adapted for defect coverage.
  Interventions: Procedure: Open Flap Debridement (OFD); Procedure: Bone Graft; Procedure: Pericardium Membrane

INTERVENTIONS:
Procedure: Open Flap Debridement (OFD) — Under Local Anesthesia , intrasulcular incisions using surgical blade #15c Then, a full thickness mucoperiosteal flap will be raised . Then, the granulation tissue in the intrabony defect will be debrided and the root will be planned using manual and ultrasonic instruments followed by saline and chlorohexidine irrigation till obtaining a healthy sound bone surface.
Procedure: Bone Graft — Bovine Xenograft material packed into the debrided defect.
Procedure: Autogenous Periosteal Pedicle Graft (PPG) — * Vertical releasing incisions will be used if necessary for better access.
  * The periosteal membrane will be separated from this flap and released with one vertical incision mesially and one horizontal incision apically . Posteriorly, the periosteum remained attached to the mucoperiosteal flap for adequate blood supply.
  * periosteal membrane will be turned over to cover this defect completely and sutured with the lingual flap with a synthetic 6-0 bioabsorbable Vicryl suture. *The soft tissue flap will be sutured with 5-0 nonabsorbable prolene suture material and a periodontal dressing was given.
  Arms: Group I (Open Flap Debridement (OFD) with autogenous Periosteal Pedicle Graft (PPG) and Bone graft).
Procedure: Pericardium Membrane — A pericardium membrane was adapted for defect coverage and sutured with the lingual flap with a synthetic 6-0 bioabsorbable Vicryl suture.
  Arms: Group II (Open Flap Debridement (OFD) with Pericardium membrane and Bone graft).

SUMMARY:
The aim of this study is to compare between autogenous PPG and Pericardium membrane in management of periodontal intrabody defects in stage III periodontitis.

DETAILED DESCRIPTION:
Periodontitis is a chronic infectious disease that causes damage to periodontal tissues. One of its consequences is alveolar bone resorption, which generates horizontal or vertical bone defects and supra- or intrabony defects, causing mobility and tooth loss.

Periodontal regeneration refers to the restoration of bone, cementum and periodontal ligament to their original levels once damaged by periodontal disease. It has been shown that periodontal regeneration can be achieved by a variety of nonsurgical and surgical procedures.

Surgical modalities of periodontal regeneration include osseous grafts, guided tissue regeneration and a combination of both , Often, a new junctional epithelium is present between the regenerated alveolar bone and the previously diseased root surface.

For intrabony defects regenerative interventions included the use of enamel matrix derivatives, bone grafts, guided tissue regeneration (GTR), and biologic modifiers to achieve regeneration.

GTR is a barrier technique used for the treatment of periodontal bone defects. Guided bone regeneration (GBR) is used to enhance bone growth of the alveolus for implant placement and around peri-implant defects.

The aim of the GTR procedure is to restore destroyed periodontal support. Indeed, the placement of a physical barrier between the surgical flap and the root surface can exclude the epithelium from the healing process and can protect the blood coagulum, promoting its adherence to the root surface .

An ideal GTR membrane should possess the following promising features: appropriate mechanical strength, biocompatibility, active osteogenic property, and antibacterial strength.

Several nonresorbable and bioabsorbable materials have been used as barrier membranes in the GTR procedure , Among these, autogenous periosteal grafts, as both free and pedicle grafts, have been proposed for the treatment of periodontal defects .

The periosteum consists of three allocated zones. The first zone predominantly comprises osteoblasts; they represent 90% of the total cell population in this layer, with collagen fibrils constituting 15% of the volume. The second zone primarily consists of fibroblasts, and endothelial cells constitute the remaining spaces. The third zone is fibrous indicating the presence of the highest amount of collagen fibers and fibroblasts. The presence of such an extensive population of osteoprogenitor cells makes it an attractive tool for periodontal regeneration .

Autogenous periosteal grafts are an attractive alternative to existing barrier membrane materials since they meet the requirements of an ideal material, and they are biologically accepted. Moreover, periosteum has the potential to stimulate osteogenesis in the bony defect area .

The advantages of using an autogenous periosteal membrane are that it requires only one surgical procedure, minimizes any undesirable tissue responses during healing and has the potential for stimulating new bone formation .

Marginal periosteal pedicle (MPP) graft was introduced by Gamal and Mail-hot as a biologic GTR membrane as an attempt to manage deep angular two- and three-wall intrabony periodontal defects.

Moreover, MPP graft was examined clinically and histologically as a biologic guided tissue membrane. Not only clinical improvement was observed but also, histologic evaluation of test samples revealed coarse-fibered woven bone filling the defect nine months following therapy in three of the 10 examined newly formed tissue samples and a homogenous layer of cementum-like tissue deposition was detected in apical root notches of such samples.

The choice of using autogenous periosteal pedicle grafts was based on their biological compatibility, high vascularity, rich and diverse cellularity, acceptable rigidity, and strong regenerative capability.

A common bioresorbable barrier membrane used in GTR is collagen membrane which is made of natural polymers. The most common natural polymers used for collagen membrane fabrication are collagen type I and type III.

Natural collagen is extracted by decellularization and removal of antigenic components from primary sources which include but are not limited to porcine skin, porcine pericardium, and bovine tendon.

Some drawbacks of using a biodegradable collagen membrane include difficulties in regulating the degradation process, limited mechanical strength, the presence of residual cross-linking agents, and the potential risk of disease transmission .

The pericardium membranes, in comparison to other collagen membranes have shown an effective crosslinking, suggesting prolonged resorption time, Various in vitro and in vivo studies have managed to prove the bio-effectiveness of these pericardium membranes in enhancing bone augmentation.

Therefore, the present study will be undertaken to assess the regenerative capacity of autogenous periosteal pedicle graft in comparison with Pericardium membrane in management of Periodontal Intrabony Defects.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes aged (25-45) years old.
* Patients who exhibit signs of (stage III) periodontitis.
* Healthy individuals and free from systemic disease that may contraindicate periodontal surgery and influence the outcome of the therapy, according to the detailed questionnaire of the dental modification of the Cornell medical index .
* Patients who have not received antibiotics or any medication for at least 6 months prior to this study.
* Patients who have not undergone any type of Surgical periodontal therapy 6 months prior to the initial examination.
* Patients able to return for multiple follow-up visits.

Exclusion Criteria:

* Pregnant and lactating females .
* Teeth with mobility greater than Grade I according to Miller classification .
* Patients with any harmful habits, like smoking or tobacco chewing.
* Unacceptable oral hygiene after the re-evaluation of phase I therapy.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Attachment Level (CAL) from Baseline to 6 Months | Baseline, 3 months, and 6 months
  The distance from the cementoenamel junction (CEJ) to the bottom of the periodontal pocket will be measured in millimeters (mm) using a UNC-15 probe. Improvement in CAL indicates periodontal healing.

SECONDARY OUTCOMES:
Change in Probing Depth (PD) from Baseline to 6 Months | Baseline, 3 months, and 6 months
  Distance from the gingival margin to the base of the pocket, measured in millimeters (mm) using a UNC-15 probe.
Change in Plaque Index (PI) from Baseline to 6 Months | Baseline, 3 months, and 6 months
  Accumulation of plaque measured as a score (0-3).
Change in Gingival Index (GI) from Baseline to 6 Months | Baseline, 3 months, and 6 months
  Gingival inflammation measured as a score (0-3)
Radiographic Bone Fill Measured by Cone Beam Computed Tomography (CBCT) from Baseline to 6 Months | Baseline and 6 months
  Measurement of intrabony defect depth in millimeters (mm) and angle in degrees(°) using CBCT at baseline and 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Khalil, professor, Study Chair — Minia University; Aya Allah k Abd El-al, Lecturer, Study Director — Minia University
Locations (1):
- Faculty of dentistry, Minia University, Minya, Minya Governorate, Egypt